CLINICAL TRIAL: NCT06047132
Title: CROSS SECTIONAL CLINICAL STUDY TO DETERMINE THE PREDICTIVE ABILITY OF A PANEL OF BIOMARKERS IN SALIVA IN HEALTHY AND PERIODONTALLY AFFECTED SUBJECTS. PILOT STUDY
Brief Title: PREDICTIVE ABILITY OF A PANEL OF BIOMARKERS IN SALIVA IN HEALTHY AND PERIODONTALLY AFFECTED SUBJECTS
Acronym: FLOE
Status: Completed | Type: Observational
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Other Study IDs: 110-110923
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-12

CONDITIONS: Periodontitis; Saliva; Biomarkers
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Periodontal health status: Categorized according to 2018 classification of periodontal diseases (Papapanou et al. 2018), including healthy, gingivitis, treated periodontitis (stable/unstable), periodontitis Stages I & II, and periodontitis Stages III and IV.
  Interventions: Diagnostic Test: Salivaru biomarkers

INTERVENTIONS:
Diagnostic Test: Salivaru biomarkers — C-reactive protein (CRP), triggering receptor expressed on myeloid cells-1 (TREM-1), interleukin (IL)-1beta, metalloproteinase (MMP)-8, IL-10, IL-6, monocyte chemoattractant protein-1 (MCP-1), Macrophage Inflammatory Protein-1 Alpha (MIP-1), interferon-gamma (IFN-gamma), osteoprotegerine (OPG), Receptor activator of nuclear factor kappa B ligand (RANKL), Tumor Necrosis Factor-Alpha (TNF-alpha)

SUMMARY:
Objective: The main aim of this cross-sectional clinical study is to evaluate the predictive ability of a panel of salivary biomarkers in determining periodontal health status.

Material and methods: In this observational, cross-sectional study patients attending consecutively to the Periodontal Postgraduate Clinic at the University Complutense of Madrid. The participants will be categorized into different periodontal health status groups based on the 2018 classification of periodontal diseases, including periodontally healthy, gingivitis, treated periodontitis (stable/unstable), and various stages of periodontitis. During the screening visit, participants will undergo a comprehensive medical examination to gather relevant health information, including age, gender, weight, height, waist circumference, and drug, alcohol, and smoking history. Additionally, clinical assessments, saliva samples and microbiological parameters will be recorded. A convenience sample of 100 subjects will be recruited for this pilot study with the objective to generate data for the multivariate predictive analysis. Data analyses: Descriptive statistics will be used to report the clinical variables and patients will be grouped according to the pre-established diagnostic categories (periodontally healthy, gingivitis, treated periodontitis patient. In order to determine the possible statistical relationship with the medical, biochemical and microbiological variables assessed, a crude bivariate analysis will first be performed by applying a mean comparison test for quantitative variables (ANOVA) and a proportion comparison test for categorical variables (Chi-square). Subsequently, those variables identified as relevant in the crude analyses will be included as confounding and/or interaction factors in a binary logistic regression model, considering the presence of periodontitis as a response variable, in order to obtain crude and adjusted OR values, together with their corresponding 95% CIs. Based on the results obtained in the biomarker analysis, a relevant statistical analysis will be performed, taking into account all the variables collected in the study

ELIGIBILITY:
Inclusion criteria:

* Adults (≥ 18-year-old)
* Being able to sign an informed consent form
* Willing to participate in this observational investigation
* Diagnosed as periodontally healthy, gingivitis, treated periodontitis patient (stable / unstable), periodontitis stages I & II, or periodontitis stages III and IV (Papapanou et al. 2023)

Exclusion criteria:

Patients fitting to all the above inclusion criteria will be excluded from the study if unable to attend to the study-related procedures or if one or more of the following systemic or local exclusion criteria will be found at any time through the study:

1. Systemic exclusion criteria

   * Un-controlled diabetes (HbA1c >7)
   * Compromised general health status (≥ASA III);
   * Drug abuse, alcohol abuse, or smoking > 10 cigarettes a day;
   * Chronic use of corticosteroids, NSAIDs, or immune modulators (any type/dose);
   * No recent Asthma, hayfever, allergies, severe intolerances
   * Mouth piercing, xerostomia
   * Pregnant or nursing women.
2. Local exclusion criteria

   * History of antibiotic intake within the last 30 days
   * History of periodontal/mucogingival surgery within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from those attending in a consecutive manner to the Periodontal Postgraduate Clinic at the University Complutense of Madrid
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Salivary biomarkers | Baseline
  Combination of C-reactive protein (CRP), triggering receptor expressed on myeloid cells-1 (TREM-1), interleukin (IL)-1beta, metalloproteinase (MMP)-8, IL-10, IL-6, monocyte chemoattractant protein-1 (MCP-1), Macrophage Inflammatory Protein-1 Alpha (MIP-1), interferon-gamma (IFN-gamma), osteoprotegerine (OPG), Receptor activator of nuclear factor kappa B ligand (RANKL), Tumor Necrosis Factor-Alpha (TNF-alpha).

SECONDARY OUTCOMES:
Age | Baseline
Gender | Baseline
Hb1Ac | Baseline
  using a point of care home use diagnostic test (A1CNow+; Bayer)
Finn-risk | Baseline
  diabetic risk questionnaire
Blood pressure | Baseline
Patient's temperature | Baseline
  digital body thermometer
Habits | Baseline
  Drug, alcohol, and smoking history
Plaque index | Baseline
  Presence/Absence
Bleeding on probing | Baseline
  Presence/Absence
Suppuration on probing | Baseline
  Presence/Absence
Probing depth | Baseline
  Distance in mm between the bottom of the pocket and the gingival margin
Recession | Baseline
  Distance in mm between the amelocemental boundary and the gingival margin
Radiographic bone loss | Baseline
  Panoramic radiograph
Microbiological analyses | Baseline
  Presence and quantity of Porphyromonas gingivalis, Aggregatibacter actinomycetemcomitans and Tannerella forsythia

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, University Complutense of Madrid (UCM), Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No